CLINICAL TRIAL: NCT05754788
Title: Identification of Gene Expression Profile Associated With Favorable Prognosis in Patients Undergoing Radical Surgery for Pancreatic and Ampullary Adenocarcinoma
Brief Title: Gene Expression Profile of Resected Pancreatic and Ampullary Adenocarcinoma at Favorable Prognosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Vincenzo Mazzaferro, Vincenzo Mazzaferro, MD PhD, University of Milan, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: 217/20
Record Dates: First submitted 2023-01-10; First posted 2023-03-06 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Resectable Pancreatic Adenocarcinoma
Keywords: resectable pancreatic adenocarcinoma; gene expression profile; RNA sequencing; prognosis of pancreatic cancer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Favorable-prognosis pancreatic adenocarcinoma: Patients experiencing favorable prognosis (defined as RFS≥60 months) following resection for pancreatic adenocarcinoma
- Unfavorable-prognosis pancreatic adenocarcinoma: Patients experiencing unfavorable prognosis (defined as RFS<12 months) following resection for pancreatic adenocarcinoma

SUMMARY:
The study aims at evaluating spatially resolved gene expression profiles of pancreatic and ampullary adenocarcinoma at favorable prognosis after surgical resection, in order to identify molecular features associated to a less aggressive biologic behavior that may benefit from upfront surgery.

DETAILED DESCRIPTION:
Despite technical improvements, surgery for pancreatic adenocarcinoma is still burdened by poor survival outcomes of only 10% at 5 years, due to very high locoregional and distant recurrence rates. In order to improve such disappointing results, several studies are now focusing on the role of neoadjuvant treatment. Recent evidence shows that neoadjuvant treatment may achieve improved intention-to-treat survival outcome, increased rates of margin-negative resections and decreased incidence of lymph node metastases. However, all surgical series report that a limited subset of patients achieve long-term survival following radical surgical resection.

After a systematic review of the available evidence on molecular profiling of pancreatic adenocarcinoma published until today the investigators have undertaken a retrospective study aimed at investigating the presence of possible genetic factors associated to a less aggressive clinical behavior. Clinical, biological and pathological features collected in a prospectively maintained database of radical surgery for pancreatic adenocarcinoma will be retrospectively reviewed together with an analysis of molecular features on surgical samples belonging to patients radically operated at the National Institute of Cancer of Milan. Such features may be used to identify those patients who may benefit from upfront surgery; in such group, vascular resections and reconstructions could be considered more liberally.

The study will consist of 2 phases:

1. A preliminary exploratory phase (group A) based on approximately 20 surgical samples of patients with surgically resected pancreatic adenocarcinoma, not treated by neoadjuvant chemotherapy, in order to evaluate the intrinsic role of tumor biology and avoid the selection of molecular features associated to treatment response. This cohort will consist of 2 groups of 10 patients each with prognostically favorable (RFS≥60 months) and unfavorable tumors (RFS<12 months), respectively. Patients from the 2 groups will be matched for clinicopathological tumor-related features. Spatially resolved transcriptomic analysis will be performed by the GeoMx Digital Spatial Profiler (DSP) (NanoString Technologies, Seattle, WA, USA) on samples of the two groups and the resulting gene expression profiles will be compared, in order to identify different patterns of gene expression in prognostically different pancreatic adenocarcinomas. Such patterns will also be compared with the TCGA database.
2. A subsequent expanded phase, based on the results of the previous exploration, will take place in case a different gene expression profile is identified. The internal validation set (group B) consists in additional 20 surgical samples associated to favorable and unfavorable prognosis (10 patients each), respectively, belonging to the same institutional series and matched for clinicopathological tumor-related features. RNA-seq analysis will be carried out on these surgical samples, aiming at confirming the results of the exploratory analysis and refine the gene expression profile. In this subset, the enrolment of patients who underwent neoadjuvant treatment will be allowed.

Due to the limited number, samples from patients affected by ampullary adenocarcinoma with favorable prognosis will be analyzed in one step and compared to matched cases with unfavorable prognosis (8 patients each, group C).

Following the identification of gene expression profiles both for pancreatic and ampullary adenocarcinoma, an external validation set will be enrolled in order to perform RNA-seq analysis on additional 60-80 surgical samples from other institutions and validate the prognostic relevance of the identified pattern in predicting a less aggressive disease course.

ELIGIBILITY:
Inclusion Criteria:

• Patients >18 years old undergoing surgical treatment with curative intent for pancreatic and ampullary adenocarcinoma between 1/1/2010 and 31/12/2017 with a regular follow-up and a RFS ≥36 months including:

* Patients with locoregional lymph node metastases found at final pathology;
* Patients with residual microscopic disease found at final pathology (R1 resections);
* Presence of minimal extra-regional disease not detected pre-operatively (nodule of carcinosis, single liver metastasis, single extra-regional lymph node) and removed with the primary tumor within the same intervention.

Exclusion Criteria:

* Patients undergoing preoperative radiotherapy/chemotherapy for borderline resectable or initially unresectable tumors converted to surgical resection;
* Patients with residual macroscopic disease after surgery (R1 resections);
* Patients with metastatic disease found at laparotomy and contraindicating surgical resection, including unknown liver metastases, peritoneal carcinomatosis, distant lymph node disease;
* Patients with unavailable follow-up or surgical samples for gene analysis.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A prospectively maintained database of patients with pancreatic and ampullary adenocarcinoma undergoing radical surgical resection from 1st Jan 2000 to 31st Dec 2017 in a single institution (HPB and liver transplantation Unit, National Institute of Cancer, Milan, Italy) will be used to identify patients at favorable and unfavorable prognosis.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Favorable-prognosis gene expression pattern | 19/09/2022-29/09/2023
  Identification of DSP gene aberrations associated to favorable prognosis (≥60-month RFS) after radical surgery for pancreatic and ampullary adenocarcinoma, through comparison of prognostically favorable and unfavorable gene expression profiles found in different tumor and microenvironment compartments.

SECONDARY OUTCOMES:
TCGA comparison | 19/09/2022-29/09/2023
  Comparison of the gene expression profile found at DSP with the TCGA database in order to confirm the clinical relevance of the identified gene expression pattern associated to prognostically favorable tumors
Clinical, biological and pathological factors | 19/09/2022-29/09/2023
  Identification of clinical, biological and pathological prognostic factors associated to favorable prognosis (≥60-month RFS) after radical surgery for pancreatic adenocarcinoma
External validation of gene expression profile | 19/09/2022-29/09/2023
  External validation of the identified gene expression profile through gene expression analysis of surgical samples from patients undergoing radical surgery for pancreatic adenocarcinoma in a different institution

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute of Milan, Milan, Italy

REFERENCES:
- [Background] Torres C, Grippo PJ. Pancreatic cancer subtypes: a roadmap for precision medicine. Ann Med. 2018 Jun;50(4):277-287. doi: 10.1080/07853890.2018.1453168. Epub 2018 Mar 22. PMID 29537309
- [Background] Pihlak R, Weaver JMJ, Valle JW, McNamara MG. Advances in Molecular Profiling and Categorisation of Pancreatic Adenocarcinoma and the Implications for Therapy. Cancers (Basel). 2018 Jan 12;10(1):17. doi: 10.3390/cancers10010017. PMID 29329208
- [Background] Silvestris N, Brunetti O, Bittoni A, Cataldo I, Corsi D, Crippa S, D'Onofrio M, Fiore M, Giommoni E, Milella M, Pezzilli R, Vasile E, Reni M. Clinical Practice Guidelines for Diagnosis, Treatment and Follow-Up of Exocrine Pancreatic Ductal Adenocarcinoma: Evidence Evaluation and Recommendations by the Italian Association of Medical Oncology (AIOM). Cancers (Basel). 2020 Jun 24;12(6):1681. doi: 10.3390/cancers12061681. PMID 32599886